CLINICAL TRIAL: NCT02623231
Title: The Effect of Escitalopram on Mood, Quality of Life and Cognitive Functioning in Glioblastoma Patients
Acronym: Cipralex&GBM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director of R & D department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0600-15
Record Dates: First submitted 2015-11-10; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: GBM; Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- escitalopram (Experimental): Group number 1 will include 50 patients, who will receive Escitalopram at a dose of 10 mg for a week exceeding 20 mg immediately after diagnosis for 3 months
  Interventions: Drug: Escitalopram; Drug: placebo
- placebo (Placebo Comparator): Group number 2 will include 50 patients, who will receive Placebo at a dose of 10 mg for a week exceeding 20 mg immediately after diagnosis for 3 months
  Interventions: Drug: Escitalopram; Drug: placebo

INTERVENTIONS:
Drug: Escitalopram — Group number 1 will include 50 patients, who will receive Escitalopram at a dose of 10 mg for a week exceeding 20 mg immediately after diagnosis for 3 months
  Other Names: Cipralex
Drug: placebo — group # 2 Will include 50 patients , who will receive placebo at a dose of 10 mg for a week exceeding 20 mg immediately after diagnosis for 3 months

SUMMARY:
Testing the effect of providing an antidepressant and anxiety-type escitalopram for patients with glioblastoma on patient's quality of life including the effect of treatment on mood and cognition during treatment.Two subgroups will fill questionnaires :

* Questionnaire mini mental state exam (mmse) which is the maximum score of 30. A score of below 24 indicates a flaw in the level of dementia
* Questionnaire depression / mood PHQ9P(Pa t i e n t H e a l t h Qu e s t i o n n a i r e - 9)
* The M. D. Anderson Symptom Inventory (MDASI)
* Evaluation of the hospital situation awareness (clinical assessment and questionnaire)
* Cognitive assessment which will be carried out by the Department neuropsychological and include:

  * Executive function (Stroop)
  * Abstract Reasoning (similarities)
  * -Auditory and Spatial Attention (Digit span, Spatial span) visual memory and remembering Literature
  * Memory function - visual and auditory (ROCF, RAVLT)
  * Language function: Naming and verbal fluency
  * Mindstreems Neurotrax

DETAILED DESCRIPTION:
This study is planned as prospective randomized, controlled, double-blind study.

Patients will undergo resection or biopsy of glioblastoma (newly diagnosed glioblastoma), will randomization ratio of 1: 1 by the pharmacist (by age,Karnofsky score, extent of tumor resection), for two research groups:

Group number 1 will include 50 patients, who will receive Escitalopram or Placebo at a dose of 10 mg for a week exceeding 20 mg immediately after diagnosis for 3 months. . The dose study is fixed and is not aimed at symptomatic treatment of anti-depressant (such as major depression).

ELIGIBILITY:
Inclusion Criteria:* men and women

* Aged 18-80
* who signed an informed consent form
* patients that underwent biopsy or resection of brain glioblastoma.
* KPS≥70
* Patients that are stable in terms of seizures who take only one antiepileptic drug

Exclusion Criteria:

* Patients who suffered from depression within five years,
* Patients treated with antidepressants
* Are not able to answer the questionnaires because of an inability to communicate
* Patients treated with inhibitors (MAOI) such as: nialamide , isocarboxazid , iproniazid, phenerzine, tranylcypromine
* Patients who suffer from epilepsy.
* Patients who suffer from Parkinson's
* Patients who suffer from cardiac dysfunction or heart attack recently.
* Patients with eye problems in expanding pupils - can result in the development of glaucoma and closed angle.
* Severe renal dysfunction. (creatinine clearance <30 mL / min). , Creatinine less than 1.5 times the upper limit of normal or end-stage renal disease
* Hepatic insufficiency -bilirubin General> 1.5 times the upper limit of normal, Hepatic Enzymes less than 2.5 times upper limit of normal
* Pregnant women
* a score of less than 24 test The mini-mental state examination (MMSE)
* allergy to any component of the drug- Talc, croscarmellose sodium, Microcrystalline Cellulose silicified, Magnesium stearate, Hypromellose, Macrogol 400, Titanium Dioxide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
changes in patients mood and cognitive function according to the neuropsychological assessment that includes patient health questionnaire (PHQ9) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grossman, MD, Principal Investigator — tasmc,
Locations (1):
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel